CLINICAL TRIAL: NCT05644847
Title: Effects of Whole Body Vibration Training on Lumbar Proprioception and Postural Stability in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/17
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Proprioception, Postural Balance

STUDY DESIGN:
Intervention Model Description: Single Blinded Parallel Randomised controlled Trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be a another person who will be unaware of the group the participant belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Core Stability Training Group) (Active Comparator): Participants in the control group/ core stability training group will be instructed to perform core stability exercises which will include pelvic bridge, straight leg bridge, modified kneeling with elbow support, and leg lifts and squats, with 60 seconds rest intervals between each activity. All these core exercises will be performed on a stable surface and will be progressed in difficulty by increasing the no. of repetitions and no. of sets weekly. Every session will be preceded by 5 minutes of warm-up and end with 5 minutes of cool-down exercises. A total of 12 sessions will be conducted over a period of 04 weeks.
  Interventions: Procedure: Core Stability Training
- Group B (Whole body Vibration Training Group) (Experimental): Participants in the dynamic WBV group will be provided with dynamic exercises along with WBV training at 50 Hz frequency.
  Participants will be instructed to perform 1-3 sets of 5-12 repetitions each of pelvic bridge, straight leg bridge, modified kneeling with elbow support, and leg lifts and squats on the WBV equipment, with a 60-second rest interval between each activity. The vibration speed and no. of sets and repetitions will be increased progressively. A total of 12 sessions will be conducted over a period of 04 weeks.
  Interventions: Other: Whole Body Vibration Training; Procedure: Core Stability Training

INTERVENTIONS:
Other: Whole Body Vibration Training — WBV training will be performed on a commercial vibrating platform (Healthmate HM01-08VF Gym Fitness Equipment Step Vibration Machine, China), which produces vertical sinusoidal vibrations. Participants in the dynamic WBV group will be provided with dynamic exercises along with WBV training. The vibration speed level will be progressed from level 5 to level 10 during the course of the treatment sessions
  Arms: Group B (Whole body Vibration Training Group)
Procedure: Core Stability Training — Core stability exercises will include pelvic bridge, straight leg bridge, modified kneeling with elbow support and leg lifts and squats, with 60 seconds rest interval between each activity. All these core exercises will be performed on a stable surface and will be progressed in difficulty by increasing the no. of repetitions and no. of sets on a weekly basis. Every session will be preceded by 5 minutes of warm-up and end with 5 minutes of cool-down exercises.

SUMMARY:
Spinal proprioception is integral for maintaining trunk stability during the performance of both static and dynamic tasks. Proprioceptive feedback contributes towards joint position sense and postural stability. Several treatment approaches are available for improving proprioception, one such modality is whole body vibration. The evidence supporting the effectiveness of WBV in improving postural stability is scarce. Moreover, the population of interest for this study is healthy adults because this age group is often neglected in the research related to balance and postural stability however incidence of falls in this age group is high as per latest evidence. The aim of this study is to compare the effect of whole-body vibration along with core stability training versus core stability training alone on lumbar proprioception and postural stability in healthy adults.

DETAILED DESCRIPTION:
Stability of the lumbar spine is required for static and dynamic functioning in daily life activities. Spinal proprioception is one of the major feedback mechanisms which contribute to spine positioning and trunk stability. Sense of proprioception is processed by the central nervous system based on the afferent information received by mechanoreceptors located in muscle spindles, Golgi tendon organs, and joint capsules. Proprioceptive feedback contributes toward joint position sense which is integral for trunk control, postural stability, and balance. Defective proprioceptive feedback can impair normal coordinated trunk motion which, in turn, can lead to decreased stability and a higher risk of musculoskeletal injury.

Several treatment approaches are available that aim to improve proprioception such as balance board, taping, bracing, manual therapy techniques, etc. However, with recent technological advancements, newer treatment modalities have been introduced that aim to improve joint position sense. One such modality is whole body vibration where the individual is exposed to mechanical vibrations through a device or a vibrating platform. It requires the individual to perform exercises on a platform vibrating between 1-50 Hz. The effects of WBV are currently being studied in the field of rehabilitation. Past research has established the neurophysiological basis of whole-body vibration on proprioception. Studies have demonstrated that training via WBV causes a continuous proprioceptive stimulation which enhances neuromuscular receptivity of the muscle spindle and helps improve muscle function. Existing literature has established the effectiveness of WBV to improve muscle strength, endurance, and power, moreover, it is also suitable for individuals who cannot perform strenuous exercise. However, there is conflicting evidence on the role of WBV on postural stability, and needs further exploration. Core strengthening is already a part of treatment regimens focused on improving trunk stability, and is backed by a vast literature. The current study is focused on comparing the effects of WBV along with core strengthening protocol verse core stability training alone in adults. If WBV is found effective, it can help in providing training protocols using WBV for improving muscle activation among untrained and enhancing performance among trained sports personnel. The main objective of this study is to compare the effect of whole-body vibration along with core stability training versus core stability training alone on lumbar joint position sense error and postural stability in healthy adults. For the purpose of this study, 42 participants meeting the inclusion criteria will be recruited. After baseline assessment participants will be randomly allocated to two groups i.e. Whole-Body Vibration along with core training and core stability training alone. Participants will receive 12 treatment sessions over the course of four weeks after which post treatment assessment of outcome measures will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults aged 18-25 years
* Both males and females willing to participate in the study
* No participation in a regular exercise or physical activity program
* Subjects with fall risk score (FRS) > 1.5 on Biodex balance system

Exclusion Criteria:

* Individuals suffering from any acute or chronic co-morbidities of musculoskeletal, neurologic, cardiovascular or systemic origin
* Subjects with history of low back pain or any vestibular disorders, inner ear infections, or hearing loss, which could affect balance and proprioception
* Pregnant females

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Lumbar Proprioception/ Lumbar Joint Position Sense Test | 04 Weeks
  Lumbar Proprioception/ Lumbar Joint Position Sense Test will be measured using inclinometer having excellent validity and reliability. Two inclinometers will be used simultaneously for measuring the flexion and extension ROM. Repositioning accuracy will be assessed with participants trying to reproduce the target position. Active repositioning error i.e. the difference between a target position and the reached position of the patient will be measured. A higher repositioning error indicates poor joint position sense or proprioception.

SECONDARY OUTCOMES:
Postural Stability | 04 Weeks
  Postural stability of participants will be assessed using Biodex balance system SD. Scores for overall stability, anteroposterior and mediolateral stability will be noted for each participant. A higher score indicates poor postural stability.

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital Department of Rehabilitation, Rawalpindi, Punjab Province, Pakistan